CLINICAL TRIAL: NCT02332447
Title: Efficacy of Naloxone in Reducing Postictal Central Respiratory Dysfunction in Patients With Epilepsy
Acronym: ENALEPSY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014-853; 2014-003003-30 (EudraCT Number)
Record Dates: First submitted 2015-01-05; First posted 2015-01-06 (Estimated); Last update posted 2025-09-26 (Actual); Status verified 2024-10

CONDITIONS: Epilepsy
Keywords: Tonic-clonic seizures; Naloxone; SUDEP
MeSH Terms: conditions — Epilepsy; Seizures; Sudden Unexpected Death in Epilepsy | interventions — Naloxone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NALOXONE (Experimental)
  Interventions: Drug: naloxone
- PLACEBO (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: naloxone — A single dose of 1 ml of naloxone (i.e 0.4 mg) or placebo will be administered by the supervising nurse or physician, using direct intravenous injection with a 5 ml syringe through peripheral venous catheter of which all patients will be equipped throughout the video-EEG.
  The evolution from a partial seizure to a GTCS being gradual, and the total duration of the seizure ranging from 2 to 3 minutes, the injection will be prepared during the course of the seizure. Given the assumptions about the role of endogenous opioids release in the spontaneous termination of seizures, naloxone will be administrated immediately after the end of the GTCS and not before. Specifically, treatment administration will be performed within the 2 minutes following the end of the GTCS.
  Arms: NALOXONE
Drug: Placebo — Placebo will be isotonic sodium chloride which preparation in 1 ml vials will be centralized by the pharmaceutical department of Edouard Herriot Hospital to ensure its indistinguishability from naloxone A single dose of 1 ml of naloxone (i.e 0.4 mg) or placebo will be administered by the supervising nurse or physician, using direct intravenous injection with a 5 ml syringe through peripheral venous catheter of which all patients will be equipped throughout the video-EEG.
  The evolution from a partial seizure to a GTCS being gradual, and the total duration of the seizure ranging from 2 to 3 minutes, the injection will be prepared during the course of the seizure. Given the assumptions about the role of endogenous opioids release in the spontaneous termination of seizures, naloxone will be administrated immediately after the end of the GTCS and not before. Specifically, treatment administration will be performed within the 2 minutes following the end of the GTCS.
  Arms: PLACEBO

SUMMARY:
Sudden unexpected death in epilepsy (SUDEP) primarily affects young adults with drug-resistant epilepsy, with an incidence of about 0.4%/year. The diagnosis of SUDEP requires that anamnestic data and post-mortem examination do not reveal a structural or toxicological cause for death. Generalized tonic-clonic seizures (GTCS) are the main risk factor for SUDEP, which they appear to trigger in most instances. Indeed, experimental and clinical data strongly suggest that most SUDEP result from a postictal respiratory dysfunction progressing to terminal apnea, later followed by cardiac arrest.

Postictal apnea could partly derive from a seizure-induced massive release of endogenous opioids. Animal studies suggest that such seizure-related release of endogenous opioid peptides participate to termination of seizures. In patients with epilepsy, functional imaging studies have confirmed that seizures induce release of endogenous opioids. The brainstem respiratory centers contain the highest density in opioid receptors, accounting for respiratory depression being one of the cardinal symptoms of opioid overdose.

The investigators hypothesis is that SUDEP partly results from a post-ictal apnea promoted by a GTCS-induced massive release of endogenous opioids, and that an opioid antagonist could represent an effective preventive treatment of SUDEP. This could be achieved by chronic administration of Naltrexone, an opioid antagonist that has been used in a large population of patients with chronic alcoholism at high risk of seizures, without showing any pro-convulsant effect. This is a crucial feasibility issue since antagonising a mechanism thought to participate to seizure termination could theoretically aggravate seizures.

Before evaluating the efficacy of chronic administration of naltrexone, it is legitimate to perform a proof of concept study by testing the acute effect of an equivalent injectable treatment (Naloxone) in the immediate aftermath of GTCS recorded inhospital during video-EEG monitoring of patients with refractory epilepsy. One third of these patients develop postictal respiratory dysfunction and hypoxemia, which should be reduced by the investigators intervention if the investigators hypothesis is correct.

The main objective of the study is to evaluate the efficacy of 0.4 mg intravenous naloxone, versus placebo, administered in the immediate aftermath of a GTCS, in reducing the severity of the postictal central respiratory dysfunction occurring after the end of the seizure, as measured by pulse oximetry.

About 25% of patients with drug-resistant partial epilepsy who undergo long-term video-EEG monitoring develop at least one partial secondary generalized tonic-clonic seizure. However, these patients cannot be individualized a priori. Therefore, all adult patients with drug-resistant epilepsy who will undergo long-term video-EEG monitoring in one of the participating centres, will lack all exclusion criteria, and will give their written informed consent to participate to the study if they develop GTCS, will be included in the study. They will all benefit from continuous monitoring of pulse oximetry (together with video, EEG, and respiration recordings), and will be equipped with a peripheral venous catheter throughout the video-EEG. The modalities of the video-EEG monitoring will be consistent with the current practices and similar across the 8 centres (apart from the venous catheter which is not standard practice).

In case of occurrence of a generalized tonic-clonic seizure, patients will be randomized (1:1) to receive intravenous naloxone (0.4 mg) or placebo. Placebo will be isotonic sodium chloride which preparation and packaging will be centralized to ensure its indistinguishability from naloxone. Randomization will be centralized and stratified by centre. The evolution from a partial seizure to a GTCS being gradual, and the total duration of the seizure ranging from 2 to 3 minutes, the injection will be prepared during the course of the seizure. Given the assumptions about the role of endogenous opioids release in the spontaneous termination of seizures, naloxone will be administrated immediately after the end of the GTCS and not before.

All digital data (video, EEG, respiration, SpO2) will be centralized and evaluated blind to other data by the PI of the study who will not be involved in the video-EEG monitoring of the included patients. The same automatic and objective analysis of SpO2 data than the one already developed in the PHRC REPOMSE will be performed.

DETAILED DESCRIPTION:
Sample size was revised using a log rank test with a two-sided alternative hypothesis. For a significance level of 5% (two-tailed), assuming a hazard ratio of 2.414 calculated, i.e based on an effect size similar to the effect size of oxygenotherapy in a delay of 60 seconds (Rheims et al., 2019), 40 events should be observed to reject the null hypothesis in 80% of cases,. A proportion of 89% of patients being expected to recover SpO2 ≥ 90% 120 seconds after the end of the seizure and considering a proportion of unusauble records for technical reasons of 20%, at least 54 patients should be randomized.

Assuming that about 10% of patients with drug-resistant partial epilepsy who undergo long-term video-EEG monitoring develop at least one partial secondary generalized tonic-clonic seizure, a total of 554 patients will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* For inclusion
* Adult patient (≥ 18 years) suffering from drug-resistant partial epilepsy
* Patient undergoing long-term video-EEG monitoring in one of the participating centre to record and characterize its seizure
* Patient who gave its written informed consent to participate to the study For randomization
* Patient who suffers a secondary generalized tonic-clonic seizure during the long-term video-EEG monitoring while being supervised by a nurse or a physician

Exclusion Criteria:

* Age < 18 years
* Patient that has already been randomized in this study
* Pregnant or breastfeeding women
* Hypersensitivity to naloxone
* History of severe heart disease (myocardial infarction, heart failure disorder, arrhythmia severe hypertension)
* Ongoing opioïd treatment, including both pure agonists and partial agonists
* Addiction to opioïds, heroin, or any similar substance
* Patient participating in another drug trial for less than 2 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 485 (Actual)
Dates: Start 2015-06-26 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Delay between the end of the seizure and recovery of oxygen saturation (SpO2) ≥ 90% | during at least 5 seconds between 30 seconds and 5 minutes after the end of the GTCS

SECONDARY OUTCOMES:
Delay between the end of the GTCS and recovery of oxygen saturation (SpO2) ≥ 90% | during at least 5 seconds between 30 seconds and 5 minutes after the end of the GTCS.

OTHER OUTCOMES:
Proportion of patients whose SpO2 is <90%, <85%, 80% and 70% during at least 5 seconds 30 seconds, 1 minute, 2 minutes, 3 minutes, 4 minutes and 5 minutes after the end of the GTCS. | during at least 5 seconds 30 seconds, 1 minute, 2 minutes, 3 minutes, 4 minutes and 5 minutes after the end of the GTCS.
Desaturation nadir between 30 seconds and 5 minutes after the end of the GTCS | between 30 seconds and 5 minutes after the end of the GTCS
Number of patients who show postictal apnea, defined as the absence of chest expansion during a period > 10 seconds between 30 seconds and 5 minutes after the end of the GTCS. | between 30 seconds and 5 minutes after the end of the GTCS.
Number of patients in whom 02 administration is required within the ten minutes following the end of a GTCS | within the ten minutes following the end of a GTCS
Number of patients in whom cardiorespiratory rescue procedure is required within the ten minutes following the end of a GTCS | Within the ten minutes following the end of a GTCS
Total duration of the postictal generalized EEG suppression, defined as lack of detectable EEG activity >10 mV in amplitude on all leads | Within the ten minutes following the end of a GTCS
Total duration of the postictal coma, defined as the delay between the end of the seizure and the recovery of consciousness assessed by the ability to meet one single verbal command (handshake). | Within the 120 minutes following the end of a GTCS
Report of adverse events observed throughout the study | 36 days
Assessment of pain, using a visual analog scale, immediately after the recovery of consciousness following the postictal coma | Within the 120 minutes following the end of a GTCS
Total duration of the postictal immobility, defined as the delay between the end of the seizure and the first spontaneous movement of the patient, as assessed on the video recording. | Within the 120 minutes following the end of a GTCS
Number of patients who have a second GCTS within 120 minutes after the intravenous injection | Within the 120 minutes following the end of a GTCS

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain RHEIMS, Doctor, Study Director — Hospices Civils de Lyon
Locations (1):
- Service de Neurologie Fonctionnelle et d'Epileptologie et Institut des Epilepsies Hôpital Neurologique, Lyon, France

REFERENCES:
- [Result] Rheims S, Valton L, Michel V, Maillard L, Navarro V, Convers P, Bartolomei F, Biraben A, Crespel A, Derambure P, de Toffol B, Hirsch E, Kahane P, Martin ML, Tourniaire D, Boulogne S, Mercier C, Roy P, Ryvlin P; ENALEPSY study group. Efficacy of naloxone in reducing postictal central respiratory dysfunction in patients with epilepsy: study protocol for a double-blind, randomized, placebo-controlled trial. Trials. 2016 Nov 3;17(1):529. doi: 10.1186/s13063-016-1653-1. PMID 27809868